CLINICAL TRIAL: NCT05012462
Title: Clinical Evaluation of the CM-1500 During Apheresis Blood Donation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zynex Monitoring Solutions (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: ZMS-1500-2021-Apheresis
Record Dates: First submitted 2021-08-06; First posted 2021-08-19 (Actual); Results first posted 2024-12-06 (Actual); Last update posted 2024-12-06 (Actual); Status verified 2024-12

CONDITIONS: Fluid Loss

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Apheresis Platelet Donation: CM-1500 (Experimental): The subjects will be connected to the CM-1500 during apheresis platelet donation
  Interventions: Device: CM-1500
- Apheresis Platelet Donation: CM-1600 (Experimental): The subjects will be connected to the CM-1600 during apheresis platelet donation
  Interventions: Device: CM-1600

INTERVENTIONS:
Device: CM-1500 — The CM-1500 is a U.S. FDA cleared non-invasive monitoring device that simultaneously monitors five (5) parameters of a patient's body. A combination of these parameters is represented by a single number known as the Relative Index value.
  Arms: Apheresis Platelet Donation: CM-1500
Device: CM-1600 — The CM-1500 is a U.S. FDA cleared non-invasive monitoring device that simultaneously monitors Bioelectrical Impedance, Photoplethysmography (PPG) Amplitude, ECG Amplitude and Skin Temperature. A combination of these parameters is represented by a single number known as the Relative Index value.
  Arms: Apheresis Platelet Donation: CM-1600

SUMMARY:
The study is a prospective, single-arm, non-randomized, non-blinded, non-controlled, non-significant risk, single center study enrolling up to 200 healthy adult subjects consented to undergo an apheresis donation procedure. Subjects will be connected to the Zynex Cardiac Monitor, Model 1500 (CM-1500) to characterize changes in the relative index during an apheresis donation procedure.

ELIGIBILITY:
Inclusion Criteria:

* Ability to provide written informed consent
* Ability and willingness to comply with the study procedures and duration requirements
* 18 years of age or older
* Consented to undergo an apheresis procedure with an automated blood component device

Exclusion Criteria:

* Females who are pregnant or breastfeeding
* Undergone an amputation of the left upper extremity
* Diagnosed with dextrocardia
* Subjects who have a pacemaker

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 77 (Actual)
Dates: Start 2021-09-20 (Actual); Primary Completion 2022-12-20 (Actual); Study Completion 2022-12-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Samantha Mack, MD, Principal Investigator — Vitalant Blood Donation
Locations (1):
- Vitalant Blood Donation, Denver, Colorado, United States

IPD SHARING:
Plan to Share IPD: No
There is not a plan to make IPD available

REFERENCES:
- See also: Related Info — http://www.zynexmonitoring.com

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Apheresis Platelet Donation: CM-1500 | Apheresis Platelet Donation: CM-1600
Started | 46 | 31
Completed | 42 | 28
Not Completed | 4 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Apheresis Platelet Donation: CM-1500 | Apheresis Platelet Donation: CM-1600 | Total
Number analyzed (Participants) | 46 | 31 | 77
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.3 (17.2) | 58.7 (12.5) | 50.7 (16.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 15 | 40
  Male | 21 | 16 | 37
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 46 | 31 | 77

OUTCOME MEASURES:

1. Primary Outcome: Characterize Changes in the Relative Index During an Apheresis Procedure
Description: The objective of the study is to characterize changes in the Relative Index (RI) as a representation of its associated parameters during apheresis. This was measured by averaging the RI values after the procedure. Changes in parameters from their baseline can be used as an indicator of potential change in fluid status. This change may be reflected in the RI since it is a summated value (weighted summation of percent change) combining the changes of the parameters into a single value. In the case of fluid loss such as apheresis the RI value may decrease as a result of changes in the parameters which can change in response to fluid status change. The RI is a unitless value with no set min. or max. Within the context of this trial trying to evaluate the RI, a decrease from 100 was considered a good outcome. However, in clinical use, the RI should not be used as an indicator of patient status, instead it could be used to monitor trending of patient parameters relative to their baseline.
Time Frame: Duration of apheresis procedure (e.g., 2 - 3hrs)
Population: 4 subjects were withdrawn from the CM-1500 Arm, and 3 subjects were withdrawn from the CM-1600 Arm
Measure: Mean (Standard Deviation); unit: Relative Index
Arm/Group | Apheresis Platelet Donation: CM-1500 | Apheresis Platelet Donation: CM-1600
Number analyzed (Participants) | 42 | 28
Relative Index | 94.9 (5.6) | 99.3 (26.3)

ADVERSE EVENTS:
Time Frame: Adverse Event data were collected during subject participation and for 24hrs following, a total of up to 29hrs.
Arm/Group | Apheresis Platelet Donation: CM-1500 | Apheresis Platelet Donation: CM-1600
All-Cause Mortality (participants affected / at risk) | 0/46 | 0/31
Serious Adverse Events (participants affected / at risk) | 0/46 | 0/31
Other Adverse Events (participants affected / at risk) | 1/46 | 1/31
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Apheresis Platelet Donation: CM-1500 (N=46) | Apheresis Platelet Donation: CM-1600 (N=31)
Skin Irritation (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) — Minor skin irritation due to adhesive backing on electrodes

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-02-28): https://cdn.clinicaltrials.gov/large-docs/62/NCT05012462/Prot_SAP_000.pdf